CLINICAL TRIAL: NCT01025583
Title: Efficacy of a New Hypotonic Oral Rehydration Solution Containing Zinc and Prebiotics in the Treatment of Children With Acute Diarrhea
Brief Title: Oral Rehydration Solution With Zinc and Prebiotics in Acute Diarrhea
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Roberto Berni Canani, Department of Pediatrics University Federico II of Naples, Italy
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 184/08; 01§/2008 (Other Grant/Funding Number: Mother and Child Health Association)
Record Dates: First submitted 2009-12-02; First posted 2009-12-03 (Estimated); Last update posted 2010-01-13 (Estimated); Status verified 2009-12

CONDITIONS: Diarrhea
Keywords: acute gastroenteritis; intestinal infection; intestinal fluid secretion; intestinal microflora; treatment of childhood acute diarrhea
MeSH Terms: conditions — Diarrhea | interventions — Prebiotics

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- group 1 (standard ORS) (Active Comparator): Children with acute diarrhea receive standard hypotonic ORS.
  Interventions: Dietary Supplement: hypotonic oral rehydration solution
- Group 2 (hypotonic super-ORS) (Active Comparator): Children with acute diarrhea receive hypotonic super-ORS containing zinc and prebiotics.
  Interventions: Dietary Supplement: Hypotonic oral rehydration solution with Zn and prebiotics

INTERVENTIONS:
Dietary Supplement: hypotonic oral rehydration solution — 30-50 ml/kg of ORS in 3-4 h for mild dehydration and with 50-100 ml/kg of ORS in 3-4 h for moderate dehydration, and to administer 10 ml/kg/die of ORS in a graduated glass or bottle for dehydration prevention until cessation of symptoms.
  Other Names: REIDRAX
  Arms: group 1 (standard ORS)
Dietary Supplement: Hypotonic oral rehydration solution with Zn and prebiotics — 30-50 ml/kg of ORS in 3-4 h for mild dehydration and with 50-100 ml/kg of ORS in 3-4 h for moderate dehydration, and to administer 10 ml/kg/die of ORS in a graduated glass or bottle for dehydration prevention until cessation of symptoms.
  Other Names: PREREID
  Arms: Group 2 (hypotonic super-ORS)

SUMMARY:
Hypotonic oral rehydration solutions (ORS) containing zinc and/or prebiotics have been proposed for the treatment of pediatric acute diarrhea but conclusive clinical data about their effect are scanty, especially for children living in developed countries. The investigators aim to evaluate the efficacy of a new hypotonic ORS containing zinc and prebiotics in children with acute diarrhea.

DETAILED DESCRIPTION:
Study Design and Funding Prospective, randomized controlled trial in collaboration with family pediatricians, who care for children up to 14 years of age in the Italian Public Health System. The study protocol was illustrated and discussed during 3 meetings. The research is not funded by any pharmaceutical company and all the authors declared no conflict of interest. The study protocol was reviewed and approved by the Ethics Committee of the University Federico II of Naples.

Participants Children 3-36 months old seen in the pediatrician offices from November 2007 to March 2008 presenting acute diarrhea lasting less than 48 h are considered eligible for the study. Exclusion criteria are: diarrhea lasting more than 48 h, malnutrition as judged by a body weight/height ratio below the 5th percentile, clinical signs of severe dehydration, clinical signs of a coexisting severe acute systemic illness (meningitis, sepsis, pneumonia), immunodeficiency, underlying severe chronic disease, malnutrition, cystic fibrosis, food allergy or other chronic gastrointestinal diseases, use of pre/probiotics in the previous 3 weeks, use of antibiotics or any antidiarrheal medication in the previous 3 weeks.

Acute diarrhea is defined as a decrease in the consistency of stools (loose or liquid) and/or an increase of frequency of evacuations (3 or >3 in 24 h), with or without fever or vomiting. Informed consent is obtained from the parents of all enrolled children. Microbiologic and other laboratory investigations performed only if required for specific clinical reasons.

Intervention Enrolled patients are randomly allocated to standard hypotonic ORS (group 1) or to super-hypotonic ORS containing zinc and prebiotics (group 2). We used two commercial ORS ORS preparations available on the market as sachets with similar cost and packaging. The composition of the two ORSs is reported in Table 1.

Randomization and Blinding Patients are allocated to each group according to a computer-generated randomization list. The researchers responsible for enrolling patients allocate the next available number upon entry into the trial. The parents are instructed to rehydrate orally their children with 30-50 ml/kg of ORS in 3-4 h for mild dehydration and with 50-100 ml/kg of ORS in 3-4 h for moderate dehydration, and to administer 10 ml/kg/die of ORS in a graduated glass or bottle for dehydration prevention until cessation of symptoms. Three to four hours after, children are fed with a normal appropriate-for-age diet including full strength lactose-containing formula or cow's milk.Treatment allocation is concealed to maintain the single-blind status. Upon enrolment, the patient's parent receive the envelope containing a written prescription of the name of the ORS product and instructions about how it should be administered. To circumvent the problems in performing a double-blind study on commercially available products in a large population, we use the third-part blind observer method to assess the efficacy of the ORS preparations. To ensure unbiased efficacy assessment, the investigators collecting the reporting forms completed by the parent are blind to the patient's treatment assignment, whereas the family pediatricians in charge of treatment allocation are excluded from efficacy assessment. The reporting forms are sent to the coordinating centre at the Department of Pediatrics for analysis. We previously used this procedure in a study of 5 probiotic preparations in children affected by acute diarrhea (Berni Canani R et al. BMJ 2007;335-340). Upon enrollment, patients undergo a physical examination and clinical history taking to identify the patient, to determine the duration and severity of diarrhea, to assess associated clinical features (fever, vomiting and dehydration) and to establish nutritional status and previous therapy. The parents of enrolled children are instructed to record daily on a specific form: i) the number of fecal outputs and their consistency; ii) the amount of daily ORS assumed by the child; and iii) possible adverse events. We also record the number of the parent's missed work days, the number of hospital admissions in each group, the use of other medications.

Outcome measures The primary outcome of the study is the rate of resolution of diarrhea 72 h after starting oral rehydration therapy. We selected this time point because of a study indicated that the risk of dehydration was highest during this period and that zinc is able to reduce diarrhea after 72 h of treatment. The latter finding was recently confirmed in a Cochrane meta-analysis.

Diarrhea is considered stopped after a patient had passed the last abnormal (loose or liquid) stools preceding a normal stool output, as applied in a previous study. Secondary outcome measures are the total amount of ORS intake in the first 24 h, the number of missed work days of the parent, the number of hospital admissions in each group, and the use of other medications. Safety was also investigated.

Sample size Fifty-seven patients in each group are required to obtain a power of the study = 80%, type 1 error = 0.05, 2-tailed test considering a difference of 25% (75% vs 50%) in the rate of resolution of diarrhea at 72 h between the study groups. This estimation is based on our preliminary data and on previous results obtained in children with acute diarrhea treated with zinc. We decide to enroll 65 patients per group considering a possible drop out up to 15%.

Statistical analysis Statistical analysis is performed by a statistician blind to individual ORS preparations received by children in the two groups. Continuous variables are expressed as means ± standard deviation (SD). For categorical variables, the Pearson chi-square test is performed. The two groups are compared for continuous variables by t-test for equality of means. After checking for assumptions, linear regression analysis with stepwise method is used to study the effect of different variables (age, sex, body weight, duration of symptoms before enrollment) on the presence of diarrhea after 72 h of treatment. Analyses are conducted on an intention-to-treat and per-protocol basis. All tests of significance are two-sided. A p value of less than 0.05 is considered significant. The statistical analysis is performed using the SPSS software package for Windows (release 16.0.0; SPSS Inc., Chicago, IL, USA) and Starts Direct (release 2.6.6).

Table 1. Composition of the two ORSs compared in the study

Standard ORS Super ORS Commercial brand name Reidrax® Prereid® Assigned group Group 1 Group 2 Osmolarity (mOsm/L) 225 200 Na+ (mmol/L) 60 50 K+ (mmol/L) 20 20 Cl- (mmol/L) 60 40 Glucose (mmol/L) 75 77 Citrate (mmol/L) 10 10 Zn2+ (mmol/L) 0 1 Fructooligosaccharides (g/L) 0 0.35 xylooligosaccharides (g/L) 0 0.35

ELIGIBILITY:
Inclusion Criteria:

* Children 3-36 months old seen in the pediatrician offices presenting acute diarrhea lasting less than 48 h are considered eligible for the study

Exclusion Criteria:

* Diarrhea lasting more than 48 h
* Malnutrition as judged by a body weight/height ratio below the 5th percentile
* Clinical signs of severe dehydration
* Clinical signs of a coexisting severe acute systemic illness (meningitis, sepsis, pneumonia)
* Immunodeficiency
* Underlying severe chronic disease
* Malnutrition
* Cystic fibrosis
* Food allergy or other chronic gastrointestinal diseases
* Use of pre/probiotics in the previous 3 weeks
* Use of antibiotics or any antidiarrheal medication in the previous 3 weeks.

Ages: 3 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 130 (Actual)
Dates: Start 2007-11; Primary Completion 2008-01 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
The primary outcome of the study is the rate of resolution of diarrhea 72 h after starting oral rehydration therapy. | From November 2007 to January 2008

SECONDARY OUTCOMES:
Secondary outcome measures are the total amount of ORS intake in the first 24 h, the number of missed work days of the parent, the number of hospital admissions in each group, and the use of other medications. | From November 2007 to January 2008

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Berni Canani, MD, PhD, Principal Investigator — Department of Pediatrics, University Federico II of Naples Italy
Locations (1):
- Pediatric Office, Naples, Italy